CLINICAL TRIAL: NCT00380198
Title: A Randomized, Double-Blind Comparison of Apadenoson and Adenosine to Treadmill Exercise Stress for Single-Photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging (MPI)
Brief Title: A Comparison Study of Apadenoson and Adenosine to Treadmill Exercise Stress.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to end program
Sponsor: Forest Laboratories (Industry)
Responsible Party: Amy Lankford, PhD, Sr. Manager, PGxHealth, LLC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: BMS068645-305; EudraCT #2006-002222-31
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Drug: Apadenoson

SUMMARY:
The purpose of this clinical research study is to compare Apadenoson and adenosine to treadmill exercise stress SPECT MPI

ELIGIBILITY:
Inclusion Criteria:

* Clinically appropriate for exercise stress testing

Exclusion Criteria:

* Contraindication to adenosine stress or inability to perform treadmill exercise test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11

PRIMARY OUTCOMES:
Agreement between MPI Summed Stress Scores for extent and severity of disease

SECONDARY OUTCOMES:
Comparison of imaging data to 6 month event data or angiography

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mittleman, MD, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (41):
  - Local Institution, Huntsville, Alabama
  - Local Institution, Santa Rosa, California
  - Local Institution, Bridgeport, Connecticut
  - Local Institution, Guilford, Connecticut
  - Local Institution, Newark, Delaware
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Gainsville, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jacksonville Beach, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Stuart, Florida
  - Local Institution, Tamarac, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Aurora, Illinois
  - Local Institution, Bannockburn, Illinois
  - Local Institution, LaGrange, Illinois
  - Local Institution, Lombard, Illinois
  - Local Institution, Winfield, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Overland Park, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Baton Rouge, Louisiana
  - Local Institution, Auburn, Maine
  - Local Institution, Westminster, Maryland
  - Local Institution, Saint Louis Park, Minnesota
  - Local Institution, Tupelo, Mississippi
  - Local Institution, Kansas City, Missouri
  - Local Institution, Albany, New York
  - Local Institution, West Islip, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Lorain, Ohio
  - Local Institution, Sandusky, Ohio
  - Local Institution, Westlake, Ohio
  - Local Institution, Wyomissing, Pennsylvania
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Johnson City, Tennessee
  - Local Institution, Houston, Texas
  - Local Institution, Richmond, Virginia
  - Local Institution, Madison, Wisconsin